CLINICAL TRIAL: NCT04349839
Title: Post-marketing Surveillance Study to Evaluate the Clinical Utility of ACRODAT in an International, Randomised, Non-interventional Study
Brief Title: ACRODAT Prospective Evaluation Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 237269
Record Dates: First submitted 2020-04-03; First posted 2020-04-16 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Acromegaly
Keywords: Insulin-like growth factor-I (IGF-I); Growth hormone (GH); Disease control
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACRODAT study arm: No intervention
  Interventions: Device: Acrodat software
- Standard Practice Arm: No intervention

INTERVENTIONS:
Device: Acrodat software — Acrodat is a newly developed software medical device to access disease activity in acromegaly based on five parameters: IGF-I, tumour size, comorbidities, symptoms and quality of life.
  Groups: ACRODAT study arm

SUMMARY:
ACRODAT® is a new software medical device developed by a group of acromegaly experts to help practising endocrinologists assess disease activity in patients with acromegaly. It uses 5 key parameters (IGF-I level, tumour status, comorbidities, symptoms and Quality of life) to evaluate the patient's health status. The purpose of this post marketing surveillance study is to prospectively evaluate whether patients monitored by ACRODAT® with appropriate clinical decisions based on disease activity status will benefit from improved treatment outcomes both in the short and in the long term.

DETAILED DESCRIPTION:
This is an international, multicentre, randomised, non-interventional, collaborative post marketing surveillance study to assess the clinical use of the newly developed software medical device named ACRODAT®. Patients newly enrolled will be followed-up over a 2 year period. Patients will be assigned to the ACRODAT® group or the Standard Practice group according to a central randomisation. Patients assigned to the ACRODAT® arm will be followed up with the treating physician using ACRODAT® at every visit. The frequency of visits will be according to standard practice in the clinic. Patients not followed up with ACRODAT® will be followed-up in accordance with the standard medical practice of the hospital where they have been recruited, until study completion (Standard Practice arm).

ELIGIBILITY:
Inclusion Criteria:

1. All patients with a confirmed diagnosis of acromegaly, aged 18 years or over, pre-treated and treatment naïve;
2. A follow-up visit is scheduled or anticipated for the patient at least once every year;
3. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of and consented to all pertinent aspects of the study.

Exclusion Criteria:

1. Patients who are surgically cured and remain controlled for at least 3 years;
2. Patients who are unable to understand the nature of the study and/or unwilling to sign an informed consent;
3. Patients who are unwilling to abide by the guidelines of the study;
4. Patients participating in any clinical trial on an investigational medicine or software medical device/evaluation tool for acromegaly.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The post marketing surveillance study population will be patients with acromegaly in specialist care clinics and hospital clinics. The results from the validation study which guided development of ACRODAT® was conducted with hypothetical patient cases which were generally described as "an adult patient with a confirmed diagnosis of acromegaly, who is presenting with the following…". Therefore, ACRODAT® may be used for all adult patients with confirmed diagnosis of acromegaly or being followed up for acromegaly.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes in IGF-I levels | 2 years
  Change from baseline in IGF-I value after 24 months of patient management based on the local lab IGF-I values ( ACRODAT® vs. standard care).
Overall disease activity score using ACRODAT® | 2 years
  Final Overall disease activity score (0-100) as measured with ACRODAT® after 24 months of patient management (ACRODAT® vs. standard care).

SECONDARY OUTCOMES:
Change in ACRODAT® score | 2 years
  Change from baseline in Overall Disease Activity Score as measured with ACRODAT® for patients in the ACRODAT® group after 24 months.
Disease activity divided in 3 categories | 2 years
  Proportion of patients in each Overall Disease Activity Category (Stable, mild Disease Activity, Significant Disease Activity) after 24 months of patient management (both groups)
Change in disease activity category | 2 years
  Change in proportions in each Overall Disease Activity Category between baseline and after 24 months of patient management in the ACRODAT® group
IGF-I normalisation at any time defined by local lab | 2 years
  Proportion of patients in each group achieving IGF-I normalisation at any time (post-baseline) during the course of the study, where IGF-I normalisation is defined as an (age adjusted) IGF-I value within the normal range defined by the local lab. This proportion will also be presented split by controlled status at baseline.
IGF-I normalisation throughout the study defined by local lab | 2 years
  Proportion of patients in each group who maintain IGF-I normalisation throughout the study, where IGF-I normalisation is defined as an IGF-I value within the normal range defined by the local lab.
IGF-I normalisation defined by local lab | 2 years
  Proportion of patients in each group achieving IGF-I normalisation at Month 24 where IGF-I normalisation is defined as an IGF-I value within the normal range defined by the local lab. This proportion will also be presented split by controlled status at baseline.
IGF-I normalisation throughout the study defined by central lab | 2 years
  Proportion of patients in each group who were 'controlled' at baseline and who maintain IGF-I normalisation throughout the study, where IGF-I normalisation is defined as an age adjusted IGF-I value within the normal range defined by the central lab. (Presented by baseline controlled status as defined by the investigator, and also by the controlled status according to the central IGF-1 lab values within the normal range).
Achieving IGF-I normalisation after 24 months defined by central lab | 2 years
  Proportion of patients in each group achieving IGF-I normalisation at Month 24 where IGF-I normalisation is defined as an age adjusted IGF-I value within the normal range defined by the central lab. This proportion will also be presented split by controlled status at baseline as defined by the baseline status by the investigator and also by the controlled status according to the central IGF-1 lab values within the normal range.
Change in IGF-I levels defined by central lab | 2 years
  Change from baseline in IGF-I defined by the central lab after 24 months of patient management. Comparison between both groups.
Disease activity on the 5 key parameters after 24 months | 2 years
  Proportion of patients with individual parameter (tumour status, IGF-I, comorbidities, symptoms, ACROQoL) ACRODAT® scores categorised as 1=Stable, 2=Mild Disease Activity, 3=Significant Disease Activity after 24 months of patient management as defined in the ACRODAT tool. Comparison between both groups
Disease activity on the 5 key parameters at all other time points then 24 months | 2 years
  Proportion of patients with individual parameter (tumour status, IGF-I, comorbidities, symptoms, ACROQoL) ACRODAT® scores categorised as 1=Stable, 2=Mild Disease Activity, 3=Significant Disease Activity at all other available time points (Month 12 at a minimum) as defined in the ACRODAT tool. For the ACRODAT® group only.
Change in disease activity category after 24 months | 2 years
  Change in proportions in each individual parameter score (i.e. 1=Stable, 2=Mild Disease Activity, 3=Significant Disease Activity) between baseline and after 24 months of patient management in the ACRODAT® group
Medical therapy at baseline | 2 years
  Proportion of patients receiving medical therapy at baseline (both groups)
Change in medical therapy | 2 years
  Proportion of patients receiving a change in medical therapy and/or change in dose at any time during the study (both groups)
Usability of the ACRODAT® tool | 2 years
  Usability of the ACRODAT® tool according to the treating physician/nurse and patient (data collected via PRAC-Test) for the ACRODAT group

CONTACTS AND LOCATIONS:
Locations (1):
- Århus University Hospital, Aarhus, Denmark